CLINICAL TRIAL: NCT06431230
Title: Dose-response Relationship and High-intensity Interval Training Effects During Physical Education Lesson on Health Markers in Adolescents
Brief Title: School-based HIIT and Dose-Response Effects
Acronym: PEER-HEART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Jaroslaw Domaradzki, PhD, Associate Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WUHSS
Record Dates: First submitted 2024-05-10; First posted 2024-05-28 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Adolescents; Physical Activity; Adipose Tissue; Blood Pressure; Cardiorespiratory Fitness
Keywords: high-intensity interval training; adolescence; body composition; resting blood pressure; responders and non-responders; dose-response
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard HIIT Experimental Group (SH-EG) (Experimental): SH-EG - Standard HIIT Experimental Group, participants who will perform typical high-intensity interval training
  Interventions: Behavioral: standard high-intensity interval training
- Standard HIIT control group (SH-CG) (No Intervention): SH-CG - Standard HIIT Control Group, participants that will not perform the HIIT cycles
- Plyometric HIIT Experimental Group (PH-EG) (Experimental): PH-EG - Plyometric HIIT Experimental Group, participants who will perform plyometric high-intensity interval training
  Interventions: Behavioral: plyometric high-intensity interval training
- Plyometric HIIT Control Group (PH-CG) (No Intervention): PH-CG - Plyometric HIIT Control Group, participants that will not perform the HIIT cycles

INTERVENTIONS:
Behavioral: standard high-intensity interval training — The project will use an intensive intermittent exercise intervention according to the high-intensity interval training programme. The programme will be implemented during physical education lessons. It involves 4 minutes of exercise in a structure of 20 seconds of intense effort and 10 seconds of rest, for a total of 8 cycles. It will be repeated twice a week (in two PE lessons) for 8 weeks. It is based on the standard physical exercises: squats, push-ups, sit-ups, toe-touches, mountain climber, jumping jacks, standing abs twist and squat to side.
  Other Names: St-HIIT
  Arms: Standard HIIT Experimental Group (SH-EG)
Behavioral: plyometric high-intensity interval training — The project will use an intensive intermittent exercise intervention according to the high-intensity interval training programme. The programme will be implemented during physical education lessons. It involves 4 minutes of exercise in a structure of 20 seconds of intense effort and 10 seconds of rest, for a total of 8 cycles. It will be repeated twice a week (in two PE lessons) for 8 weeks. However, there is a difference, comparing to the St-HIIT, related to different exercises used in protocol. This kind of HIIT programme will be based on plyometric exercises: jumping jacks, skip A, skip C, jumps back into a push-up position and returns to the squat position, throwing the legs out of support and jumping out, jumping out of a squat.
  Other Names: Pl-HIIT
  Arms: Plyometric HIIT Experimental Group (PH-EG)

SUMMARY:
There are experimental evidences of the importance of high intensity exercises in health outcomes improvement. However, there are limited knowledge about possibility to affect health outcomes in adolescents through exercises programs introduced into physical education (PE) lesson. Moreover, there is lack of the studies identifying people who do not respond to stimuli, as well as examining potential determinants of non-responsiveness. Thirdly, there are no studies examining the modification of exercise dose that should be reflected in the response in such individuals.

Aim of this human experiment is to examine the effects of one cycle of 8-weeks high-intensity interval training (HIIT) implemented in physical education lesson on: (1) body composition (proportions of the body fat to the body muscles), (2) resting blood pressure, (3) physical efficiency.

Study are conducted for two years (two cycles). Each year 300 students of two secondary schools, are involved in project: 15-16-year-olds in first year, 18-19-year-olds in second year. Students are divided in experimental groups -performing 8-weeks (twice a week) cycle of HIIT implemented into PE lesson, and the control groups - students following a typical PE programme. Each cycle consists of two parts. First part is related to the 8 weeks of HIIT training, while second part is related to the dose-expose study.

All participants are examined during project before (Pre), after (Post) and Follow-Up intervention. Second part is planned after a break of several months. Persons who do not respond to the exercise stimulus in the first part will follow individually modified programmes. They will be measured before and after this additional training.

To examine the assumed HIIT-induced changes in participants the investigators will apply: (1) anthropometric measurements: body height and weight, and BMI will be calculated, (2) body mass composition (fat and muscle mass), (3) resting blood pressure, (4) beep test which is field motor specific test to assess physical efficiency.

The results of this project will help to answer the fundamental questions about HIIT induced morphological and physiological effects in adolescents, what is important from scientific and public health point of view. Particularly, in view of the growing pandemic of obesity, common elevated blood pressure and steadily declining physical fitness in children and adolescents.

DETAILED DESCRIPTION:
I. Background Prevalence of overweight and obesity is well documented in the literature. This applies to both adults and the elderly, but increasingly also to children and school-age youth. Similar to adipose tissue, there is a constant increase in the percentage of young individuals with elevated blood pressure. Moreover, children and adolescents are steadily decreasing their physical efficiency. All these characteristics serve as indicators of overall health, defined as health-related fitness (HRF). Measurements represent the health potential that adolescents bring into adulthood, what is closely related to their efficient functioning in family and professional life.

In the battle against lifestyle diseases during adolescence, there is a growing trend towards implementing intense short-term efforts. Evidence from numerous studies confirms the effectiveness of High-Intensity Interval Training (HIIT) in reducing body weight, improving body mass index (BMI), reducing body fat, and lowering resting blood pressure. Due to the reluctance of children and adolescents to engage in physical activity during leisure time, there is an increasing systemic implementation of HIIT in physical education classes to ensure widespread physical exercise among students.

A separate issue is the lack of response to exercise in some individuals (so-called non-responders). There are few studies that attempt to find the optimal exercise dose to elicit a response in as many participants as possible, ideally in all participants (dose-response relationship). However, the effectiveness of training based on the duration of exercise and rest intervals, the type of exercises (endurance, resistance, etc.), and exercise intensity is still unknown.

II. Research Project Objectives

Therefore, the aims of this research are twofold:

1. to investigate the effectiveness of different forms of short-term, intense interval exercise in reducing body fat and resting blood pressure, as well as improving aerobic and anaerobic physical endurance;
2. after identifying non-responders and applying dose-response procedures, to develop modifications to the standard HIIT program and verify the effectiveness of these modifications in inducing the aforementioned positive changes.

Hypothesis 1. The high-intensity intervention training, practising systematically during regular physical activity lessons, will affect body composition reducing body fat (through increased fat oxidation processes from very intensive exercises) and improve the fat to muscle mass proportions. In the experimental group participants with elevated blood pressure, blood pressure improvements will be observed what is connected with several physiological cardiovascular reactions. Thirdly, intensive physical short-time interval training will improve cardiorespiratory fitness.

Hypothesis 2. There are frequency of participants who will not gain in different outcomes from intervention programme.

Hypothesis 3. Programs of the HIIT intervention, individually tailored for non-responsive persons, including different determinants, induce the expected changes in the above-mentioned outcomes.

III. Research design and work plan This project is longitudinal, planned for two years of study. Both years, called cycles, are Cluster Randomised Trials (in other words - Group-Randomized Trials, where research participants are not allocated to intervention independently, but as a group.

Each cycle of the study has two parts. First part (called Common-HIIT) has two arms: experimental and control, while second part (called Dose-Response) has four arms: two experimental and two control.

Simple random sampling without replacement is used to classify classes as experimental and control. The sampling frame is the list of classes with identifiers specific for each school (e.g. 1a, 1b, 2a etc.). Randomization process is carried out by the investigators of this study using specific library in R language.

The project enrolls two types of students groups: experimental (EG) - circa 4 classes in each school, and control (CG) - circa 4 classes in each school. In Common-HIIT part, EG perform physical training intervention, while CG take part only in typical PE lessons. In Dose-Response part, non-responders (identified as persons who will not gain the effects during first part) will be randomly (the same procedure like in first part) divided into experimental group (NRs-E) and control group (NRs-C), while responders (identified as persons who will gain the effects during first part) will also be randomly (the same procedure like in the firs part) divided into experimental (Rs-E) and control (Rs-C) group.

In Common-HIIT part, all participants are examined during preintervention, postintervention and follow-up measurements. While, in Dose-Response part they are examined twice: preintervention and postintervention dose-response intervention.

IV. Research methodology IV.1 Subject characteristics. The sample size was calculated based on pilot studies using G*Power v. 3.1, resulting in a minimum sample size of 310 individuals (with a 5% dropout margin). The study involves students from first and fourth grades, who are involved in project in first and second cycle, respectively. Two high schools in the city of Wrocław were selected for the study. Participants are separated in sex groups, what is related to rules of the schools.

IV.2. Intervention procedures. The design used a parallel group study scheme (2 schools) with three replicates. In each school a different form of intervention based generally on the principles of the HIIT programme will be implemented. In one school a classical variant is planned, while in the other a variant using a plyometric mechanism is planned.

The project use an intensive intermittent exercise intervention. In one school, a standard programme is planned, in the other a modification involving a plyometric form of exercise. The chosen high-intensity interval programme is very useful in the school setting due to its simplicity of implementation and short time. It can be easily implemented into a lesson without strongly interfering with the flow of the lesson and the fulfilment of the teacher's curricular tasks. In the intervention, 8 series of 20-second exercises and a 10-second rest are performed.

The total duration is 4 minutes.The key is to perform the exercise on an intensity of 90%-100% of maximum effort. The short duration and the possibility to use different forms of exercise makes it attractive in the opinion of the participants and has a positive effect on motivation to exercise. In the first part of the study, regardless of the forms of exercise implemented in both schools, a standard HIIT intervention programme will be used. The intervention part will be preceded by a standard 10-minute pre-session warm-up. Participants will then embark on the main programme and perform intense work lasting 20 seconds and a 10-second rest interval. In the first four weeks, they will perform between four and six series, with the aim of doing a full cycle of eight series in the following four weeks. After all the series in a given cycle have been completed, there will be a 5-minute rest period. The teacher will then move on to the planned lesson tasks derived from the core curriculum.

Achieving the correct exercise intensity is a critical factor in HIIT-type interventions. However, given that the intervention will take place in a school setting, it was assumed that participants would maintain an effort of at least 80% HRmax, throughout the 8-week period. Heart rate will be measured with Polar Verity Sense wristbands. Teacher are real-time control and motivate the student's effort as the intensity decreases.

In the second part of the research, intervention modifications will be introduced that change the stimulus doses of the programmes. The details of the design of these modifications will be derived from the results obtained from the first part of the research.The following will be modified the proportions of work and rest breaks, the structure and/or form of the exercises. Non-responsive individuals (who did not responded to the exercise in the first part by lowering their body fat and/or blood pressure and/or improving their physical performance) and those who fail to maintain an effect over a period of 8 weeks will be allocated to subgroups in which they will be trained according to an appropriate modification. to subgroups where training will be modified accordingly.

Heart rate values forming a time series will be stored in the application and exported to a database at the end of the project. These results will be collated with the measurements and survey data and used for detailed analyses.

IV. 3. Measurements. Measurements are planned in three areas: morphological, cardiovascular and physical performance. Measurements of basic morphological characteristics will be carried out. Body height will be measured using an anthropometer with an accuracy of 0.1 cm (GPM Anthropological Instruments). Body weight will be measured on an electronic scale (body composition device) with an accuracy of 0.1 kg. Body composition will be also measured. Body composition device uses bioelectrical impedance method. Fat mass, muscle mass and water will be measured. On the basis of the measured morphological characteristics and body composition, the following are calculated indicators: relative body mass (BMI), relative fat mass (FMI), relative muscle mass (SMI) and muscle to fat ratio (MMI), muscle to fat ratio (MFR).

Haemodynamic features of the blood circulation will be determined by resting measurements of systolic and diastolic blood pressure and heart rate. An electronic upper arm blood pressure monitor will be used. For the measurement of aerobic and anaerobic physical capacity, population tests are foreseen (respectively, a multi-level shuttle run, the so-called beep test.

The measurements will be supplemented by the collection of survey data. This data will be the accompanying variables in the detailed, in-depth analyses. The following surveys are planned: the economic and social situation of the pupils' families (FAS scale), physical activity (IPAQ long form questionnaire) and frequency of food intake (KomPAN questionnaire). In addition, after each lesson unit, students will complete questionnaires with the subjective feeling of fatigue scale (RPE) and the lesson attractiveness scale (PACES).

V. Statistical analysis Distributions of the collected data will be assessed. Depending on the type of distribution, parametric and non-parametric methods will be applied. In multivariate exploratory procedures, data not meeting the condition of normality of distribution will be transformed and scaled. Comparisons between multiple groups with repeated measures (MANOVA/ANOVA of mixed effects), examination of correlations (regression analysis in mixed models), examination of similarities (cluster analyses) and co-occurrence (correspondence analyses) are assumed.

For dose-response relationship analyses, it is planned to use simple linear regression, polynomial regression (2nd and 3rd degree polynomial) and various multiple comparison procedures (Multiple Comparison Procedures family).

The calculation will be carried out in the R environment [43] and other statistical software.

ELIGIBILITY:
Inclusion Criteria:

* For all participants:

  1. active student of school enrolled in project,
  2. age 14-16 or 18-20,
  3. active student of 1st class in the school (for participants 14-16 years of age) or 4th class in the school (for participants 18-20 years of age),
  4. active participation in PE lessons (no medical or other exemption from lessons),
  5. no medical contraindications
  6. signed informed consent (parent/legal guardian) in case of under-age participant).

     Exclusion Criteria:
* For all participants:

  1. commitment to structured sports training
  2. injury less than 3 months prior to the intervention

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
body fat weight (BF) | Pre-HIIT, up to 24 weeks
  tthe body composition measurement with electronic bio-impedance tool (InBody); this measurement is to evaluate the potential of the intervention in body fat reduction
skeletal body muscle mass (SMM) | Pre-HIIT, up to 24 weeks
  the body composition measurement with electronic bio-impedance tool (InBody); this measurement is to evaluate the potential of the intervention in muscle mass increase
systolic blood pressure (SBP) | Pre-HIIT, up to 24 weeks
  resting blood pressure parameter, this measurement is to evaluate the potential effect of the intervention on blood pressure, particularly the the potential to reduce resting blood pressure in people with raised blood pressure (prehypertension)
diastolic blood pressure (DBP) | Pre-HIIT, up to 24 weeks
  resting blood pressure parameter, this measurement is to evaluate the potential effect of the intervention on blood pressure, particularly the the potential to reduce resting blood pressure in people with raised blood pressure (prehypertension)
physical efficiency (CRF) | Pre-HIIT, up to 24 weeks
  cardiorespiratory fitness (CRF), evaluate the potential effect of intervention on aerobic capacity; CRF is assessed with Multistage Fitness Test (MFT), and evaluates maximum rate of oxygen intake (VO2max).
  Participants perform continuous 20-metre shuttle runs, with the individual having to reach the opposite end of the 20-metre grid before the next sound signal. The time between signals decreases with each minute, forcing individuals to increase their running speed. Initial running velocity is of 8.5 km/hr and increases the speed by 0.5 km/hr each minute thereafter. The test is comprised of 23 levels.
  The result the participant achieved (the speed on the last level before the end) is transformed and the final outcome is maximum rate of oxygen intake. However, VO2max is calculated from formula: VO₂ max = -27.4 + 6.0 (speed); where speed is determined by the level achieved by the participant before he/she is withdrawn from the test.

SECONDARY OUTCOMES:
body height (BH) | Pre-HIIT,up to 24 weeks
  measurement from basis to vertex (top of head)
body weight (BW) | Pre-HIIT, up to 24 weeks
  measurement of the body mass with InBody electronic scale
body water (BWat) | Pre-HIIT, up to 24 weeks
  the body composition measurement with bio-impedance electronic tool (InBody); this measurement is to evaluate the potential intervention risk of dehydration
sitting height (SBH) | Pre-HIIT, up to 24 weeks
  measurement from seat surface to vertex (top of head)
social-economic situation | Pre-HIIT
  Family Affluence Scale (FAS) questionnaire related to the family social-economic situation, information will be used as confounding/covariate variable Family Affluence Scale (FAS) is a tool for analysing social inequalities in health.
  It consists of six questions relating to: the student's own room by the student, number of cars in the family, number of computers in the family, trips abroad with the family for holidays or holidays, and the number of bathrooms in the house and the provision of a dishwasher with a dishwasher.
  The FAS scale takes a range from 0 to 13 points. According to international recommendations, families are divided into: poor (0-6 points); average (7-9 points) and affluent (10-13 points).
physical activity | Pre-HIIT
  International Physical Activity Questionnaire (IPAQ) related to the physical activity, The IPAQ asks about domains: leisure time, domestic and gardening-yard, work-related and transport-related activity and sitting (inactivity). Intensity of the activity is defined as: walking, moderate-intensity and vigorous intensity.
  Result can be presented as continuous scores (metabolic equivalent in minutes per week) or categorical:
  1. inactive - individuals who not meet criteria for Categories 2 or 3,
  2. minimally active - any one of the following 3 criteria:
     * 3 or more days of vigorous activity, OR
     * 5 or more days of moderate-intensity activity OR
     * 5 or more days of any combination of walking, moderate-intensity or vigorous intensity (600 metabolic equivalent-min/week).
  3. health - at least 1.5 hour of being active throughout the day
dietary intake | Pre-HIIT
  questionnaire (questionnaire of eating behaviors KomPAN) is a tool for measurement of frequency of eating specific groups of meal, it is useful for evaluation of the eating behaviors; information will be used as confounding/covariate variable
  It consists:
  1. question on the number of meals per day,
  2. follow-up questions,
  3. questions on the frequency of food intake, which are components of: index of a healthy diet (positive HDI) and unhealthy diet index (negative HDI),
  4. questions about the respondent's lifestyle and personal data (all). Answers are transform to the scores related to healthy and unhealthy dietary behaviors.
  Minimum points for both indexes is 0, maximum is 100. Scores can be transform to the categories:
  1. small intensity of traits nutrition - 0-33 points
  2. moderate intensity of traits nutrition - 34-66 points
  3. high intensity of traits nutrition - 67-100 points
fatigue perception | within 10 minutes after each cycle of HIIT
  Rating of Perceived Exertion scale (RPE) of subjectively perceived fatigue; information will be used as confounding/covariate variable It runs from 0 - 10, using numbers to rate how much effort an activity takes. It examines 4 factors: (a) how fast is breathing, (b) how fast heart is beating, (c) how tired muscles are, (d) how much is sweating.
  The RPE scale rates exertion from a scale of 6 (no exertion) to 20 (maximum effort).
  Scale:
  6 - no exertion, 7-8 - extremely light, 9-10 - very light, 11-12 - light, 13-14 - somewhat hard, 15-16 - hard (heavy) 17-18 - very hard, 19 - extremely hard 20 - maximum exertion.
perceived attractiveness of lessons | within 10 minutes after each cycle of HIIT
  Physical Activity Enjoyment Scale (PACES), the attractiveness perceived during exercise by participants; it will be used as confounding/covariate variable It contains 18 items used to assess enjoyment, particularly during the physical activity.
  Respondents are asked to rate feelings at the moment about the physical activity, using a 7-point bipolar rating scale. Eleven items are reverse scored.
  An overall enjoyment for physical activity score is determined by summing the items, with a range of 18-126 being possible.
  Higher scores indicate higher enjoyment.

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław Domaradzki, PhD, Principal Investigator — Wroclaw University of Health and Sport Sciences
Locations (1):
- Wroclaw University of Health and Sport Sciences, Wroclaw, Dolny Śląsk, Poland

IPD SHARING:
Plan to Share IPD: No